CLINICAL TRIAL: NCT06145932
Title: the Effects of Repetitive Transcranial Magnetic Stimulation and Mechanisms in Clinical Function of Essential Tremor
Brief Title: Repetitive Transcranial Magnetic Stimulation Therapy in Essential Tremor
Acronym: rTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chun-Feng Liu, Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JD-LK2023096-IR01
Record Dates: First submitted 2023-11-12; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Transcranial magnetic stimulation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS treatment group (Experimental): treated with real rTMS 1800 pulses / day,for 10 days
  Interventions: Device: real rTMS
- Sham rTMS treatment group (Sham Comparator): treated with sham rTMS 1800 pulses / day,for 10 days
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: real rTMS — treated with 1HZ rTMS 1800 pulses / day,for 10 days
  Arms: rTMS treatment group
Device: sham rTMS — treated with sham rTMS 1800 pulses / day,for 10 days
  Arms: Sham rTMS treatment group

SUMMARY:
The purpose of this study is to evaluate the efficacy and electrophysiology of repetitive transcranial magnetic stimulation in the treatment of essential tremor.

DETAILED DESCRIPTION:
This is a randomized controlled study.The purpose is to evaluate the efficacy of repetitive transcranial magnetic stimulation(rTMS) in the treatment of essential tremor,and explore the possible mechanism by detecting the changes of clinical scale and TMS-electroencephalogram(TMS-EEG), so as to seek an effective therapy for essential tremor.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as essential tremor conforming to the diagnostic criteria for essential tremor in the tremor group of the International Parkinson's and Movement Disorders Society (IPMDS).
2. Signed informed consent form.

Exclusion Criteria:

1. Complicated with brain organic diseases, epilepsy, other mental diseases, family history of dementia, metal devices implanted in the body and any contraindications to TMS;
2. History of craniocerebral surgery;
3. TMS cannot cooperate;
4. TMS-EEG examination artifacts are obvious, or cannot be analyzed due to other technical reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the treatment on the essential tremor evaluated by Essential Tremor Rating Assessment Scale (TETRAS) score | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  The TETRAS is widely used tremor evaluation scale.TETRAS has been used for evaluation tremor in patients with essential tremor focuses primarily on the assessment of activities of daily living and tremor.The TETRAS score ranges from 0 to 112. The higher the TETRAS score, the more severe the symptoms.
Changes from baseline in tremor analysis | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  This outcome reflects quantitative changes in the patient's tremor.

SECONDARY OUTCOMES:
Changes from baseline in TMS-EEG | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  Amplitudes of various frequency bands in each cortical region of TMS-EEG reflects change in the patient's brain network.
Change in Non-Motor Symptoms Rating Scale (NMSS) score from baseline | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  This outcome reflects the efficacy of non-motor symptoms. NMSS is a widely used non-motor symptom rating scale that includes 9 domains, The NMSS score ranges from 0 to 360，with higher scores associated with more severe symptoms.
Change in Mini-Mental State Examination (MMSE) score from baseline | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  The MMSE is widely used to assess cognition. The MMSE score ranges from 0 to 30. The higher the MMSE score is, the better the cognitive function is.
Change in Montreal Cognitive Assessment (MOCA) score from baseline | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  MoCA is widely used to assess cognitive abilities. MOCA scores range from 0 to 30. The higher the MOCA score, the better the cognitive function.
Changes from baseline in Hamilton Anxiety Scale(HAMA) score | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  The Hamilton Anxiety Scale(HAMA) is a widely used interview scale to measure the severity of a patient's anxiety.The HAMA score can range from 0 to 56. The higher the HAMA score is, the worse the symptoms are.
Changes from baseline in Hamilton Depression Scale-24(HAMD-24) score | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  The Hamilton Depression Scale-24(HAMD-24) is a test measuring the severity of depressive symptoms in individuals. The HAMA score can range from 0 to 56. The higher the HAMA score is, the worse the symptoms are.
Quality of Life Questionnaire (QUEST) score change from baseline | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  This outcome reflects the patient's quality of life. QUEST scores range from 0 to 120.
  The higher the QUEST score, the more severe the symptoms.
Change in Pittsburgh Sleep Quality Index (PSQI) score from baseline | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  PSQI is widely used to measure sleep quality. PSQI scores range from 0 to 21. The higher the PSQI score, The worse the quality of sleep.
Change in Fatigue Severity Scale (FSS) score from baseline | visit 1(baseline), visit 2(Day 10), visit 3(Day 30)
  FSS is widely used in the assessment of fatigue. Indicates a health problem associated with fatigue. The higher the score, the worse the fatigue
RBD Screening Questionnaire (RBDSQ) score | visit 1(baseline)
  There are 10 questions in total, including the content of dreams, the relationship between dreams and behavior, injuries and neurological diseases, etc. The total score is 0-13 points, and a score of 5 or above is considered abnormal.
Test the sleep characteristics by polysomnography (PSG) | visit 1(baseline)
  This outcome reflects the patient's sleep characteristics and to analyze specific events.
test the characteristics of vestibular evoked myogenic potential (VEMP) | visit 1(baseline)
  This is a commonly used clinical test that includes cervical vestibular evoked myogenic potential (cvemp) and ocular vestibular evoked myogenic potential (oVEPM) to assess a patient's brainstem pathways.
test the gene's type of the notch2nlc | visit 1(baseline)
  This outcome reflects the genetic diagnosis characteristics of the patient and is helpful for accurate clinical diagnosis and classification

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gironell A, Kulisevsky J, Lorenzo J, Barbanoj M, Pascual-Sedano B, Otermin P. Transcranial magnetic stimulation of the cerebellum in essential tremor: a controlled study. Arch Neurol. 2002 Mar;59(3):413-7. doi: 10.1001/archneur.59.3.413. PMID 11890845
- [Background] Lv Y, Wang M, Yang J, Shi J, Xuan T, Zhang J, Du D, Cheng J, Li H. Cerebellar repetitive transcranial magnetic stimulation versus propranolol for essential tremor. Brain Behav. 2023 Mar;13(3):e2926. doi: 10.1002/brb3.2926. Epub 2023 Feb 17. PMID 36806734
- [Background] Louis ED, Ferreira JJ. How common is the most common adult movement disorder? Update on the worldwide prevalence of essential tremor. Mov Disord. 2010 Apr 15;25(5):534-41. doi: 10.1002/mds.22838. PMID 20175185
- [Background] Louis ED. The Roles of Age and Aging in Essential Tremor: An Epidemiological Perspective. Neuroepidemiology. 2019;52(1-2):111-118. doi: 10.1159/000492831. Epub 2019 Jan 9. PMID 30625472
- [Background] Bal N, Sengul Y, Behmen MB, Powell A, Louis ED. Vestibular reflexes in essential tremor: abnormalities of ocular and cervical vestibular-evoked myogenic potentials are associated with the cerebellum and brainstem involvement. J Neural Transm (Vienna). 2023 Dec;130(12):1553-1559. doi: 10.1007/s00702-023-02652-3. Epub 2023 May 18. PMID 37199795
- [Background] Berkiten G, Tutar B, Atar S, Kumral TL, Salturk Z, Akan O, Sari H, Onaran O, Biltekin Tuna O, Uyar Y. Assessment of the Clinical Use of Vestibular Evoked Myogenic Potentials and the Video Head Impulse Test in the Diagnosis of Early-Stage Parkinson's Disease. Ann Otol Rhinol Laryngol. 2023 Jan;132(1):41-49. doi: 10.1177/00034894211067838. Epub 2022 Feb 3. PMID 35114808
- [Background] Bayramoglu B, Emre U, Erdal Y, Demirhan H, Yasak I, Yalin OO. Cervical vestibular-evoked myogenic potentials in patients with essential tremor. J Clin Neurosci. 2021 Sep;91:365-368. doi: 10.1016/j.jocn.2021.07.015. Epub 2021 Jul 30. PMID 34373053
- [Background] Jimenez-Jimenez FJ, Alonso-Navarro H, Garcia-Martin E, Agundez JAG. Sleep disorders in essential tremor: systematic review and meta-analysis. Sleep. 2020 Sep 14;43(9):zsaa039. doi: 10.1093/sleep/zsaa039. PMID 32163585
- [Background] Bugalho P, Salavisa M, Borbinha C, Fernandes M, Meira B, Barbosa R, Mendonca M. REM sleep behaviour disorder in essential tremor: A polysomnographic study. J Sleep Res. 2021 Apr;30(2):e13050. doi: 10.1111/jsr.13050. Epub 2020 Apr 23. PMID 32323893
- [Background] Rekik A, Nasri A, Mrabet S, Gharbi A, Souissi A, Gargouri A, Kacem I, Gouider R. Non-motor features of essential tremor with midline distribution. Neurol Sci. 2022 Oct;43(10):5917-5925. doi: 10.1007/s10072-022-06262-x. Epub 2022 Jul 18. PMID 35849198